CLINICAL TRIAL: NCT01726010
Title: Endoscopic Ultrasound Guided Biopsy of Subepithelial Tumors of the Upper Gastrointestinal Tract Using the 22-G-Procore Needle
Brief Title: 22-G-Procore Needle for the Diagnosis of SETs of the Upper GI Tract
Acronym: PRO-SET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 102012
Record Dates: First submitted 2012-11-04; First posted 2012-11-14 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-09

CONDITIONS: Subepithelial Tumors of the Upper Gastrointestinal Tract

ARMS (1):
- 22-G Procore Needle (Experimental)
  Interventions: Device: 22-G Procore Needle

INTERVENTIONS:
Device: 22-G Procore Needle

SUMMARY:
The goal of this prospective study is to evaluate the feasibility of the 22-G Core Biopsy Needle with reverse bevel (Procore TM) in biopsy sampling of subepithelial tumors of the upper gastrointestinal tract.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age 18 years and older
2. All patients with subepithelial tumors of the upper GI tract (maximum size: 3 cm)

Exclusion Criteria:

1. Unable to obtain informed consent
2. ASA class 4 or 5
3. known pregnancy
4. contraindication endoscopy
5. contraindication for taking biopsies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-08 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
diagnostic yield | 6 months
  Number of patients with adequate tissue sample (which allows definitive diagnosis)

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum rechts der Isar, München, Bavaria, Germany